CLINICAL TRIAL: NCT06507774
Title: The Development and Study of a 3D-Printed Model for Surgical Planning of Lung Cancer with Realistic Subsegmental Boundaries and Complete Tissue Structures
Status: Completed | Type: Observational
Sponsor: Ke Zhang (Other)
Responsible Party: Sponsor-Investigator, Ke Zhang, M.D., Affiliated Hospital of Hebei University
Organization: Affiliated Hospital of Hebei University (Other)
Other Study IDs: 19277731D
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 3D reconstruction: Patients in this group underwent surgical planning with the aid of 3D reconstruction technology, which included preoperative imaging and 3D modeling to assist in the planning of thoracic surgery.
  Interventions: Device: 3D Reconstruction Technology
- Non-3D reconstruction: Patients in this group underwent traditional surgical planning without the use of 3D reconstruction technology, relying on standard preoperative imaging and planning techniques.
  Interventions: Device: No 3D reconstruction is used

INTERVENTIONS:
Device: 3D Reconstruction Technology — Utilization of 3D reconstruction technology to assist in preoperative planning and surgical procedures for thoracic surgery patients.
  Groups: 3D reconstruction
Device: No 3D reconstruction is used — This group did not use 3D reconstruction for surgical navigation
  Groups: Non-3D reconstruction

SUMMARY:
This project focuses on the development of a precision multi-organ surgical planning model aided by artificial intelligence (AI), computer-aided design (CAD), multi-material 3D printing, and multimodal 3D modeling. The integration of these advanced technologies aims to enhance the accuracy and efficiency of preoperative planning for complex surgical procedures involving multiple organs. By leveraging AI and CAD, the project seeks to create detailed, patient-specific 3D models that incorporate various imaging modalities. These models will be used to guide multi-material 3D printing, producing highly accurate replicas of anatomical structures. The ultimate goal is to improve surgical outcomes by providing surgeons with precise and comprehensive tools for planning and executing intricate surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lung cancer
* Complete clinical case data;
* All patients underwent surgical treatment;
* Voluntarily participate in the study and sign the informed consent.

Exclusion Criteria:

* Severe comorbidities, such as uncontrolled heart disease or diabetes
* History of major surgeries or other interventions
* Unwillingness to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes all lung cancer patients who underwent surgery at the Affiliated Hospital of Hebei University from 2020 to 2023.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Operation Time | During the surgery
  Measure the total duration of the surgery in minutes.
Blood Loss | During the surgery
  Assess the total blood loss during surgery in milliliters.
Postoperative Complications | Within 30 days post-surgery
  Record any complications within 30 days post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Hebei University, Baoding, Hebei, China

IPD SHARING:
Plan to Share IPD: No